CLINICAL TRIAL: NCT01272687
Title: Epidemiological Study to Determine Mutations in the Gaucher Gene in Patients With Idiopathic Parkinson's Disease for Phenotype-genotype Correlation
Brief Title: Study to Determine Mutations in the Gaucher Gene in Patients With Idiopathic Parkinson's Disease for Phenotype-genotype Correlation
Acronym: PadGau
Status: Completed | Type: Observational
Sponsor: CENTOGENE GmbH Rostock (Industry)
Responsible Party: Sponsor
Other Study IDs: PD02/2011
Record Dates: First submitted 2011-01-07; First posted 2011-01-10 (Estimated); Last update posted 2021-04-09 (Actual); Status verified 2020-04

CONDITIONS: Parkinson Disease; Idiopathic Parkinson Disease
Keywords: Parkinson Disease; Parkinsonian Disorders; Brain Diseases; Central Nervous System Diseases; Nervous System Diseases; Neurodegenerative Diseases
MeSH Terms: conditions — Parkinson Disease; Parkinsonian Disorders; Brain Diseases; Central Nervous System Diseases; Nervous System Diseases; Neurodegenerative Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Observation: Adults (>18 years) with a confirmed diagnosis of Parkinson's disease

SUMMARY:
The genotype-phenotype correlation in patients with Parkinson's disease with specific mutations in the glucocerebrosidase gene (Gaucher gene) is known from own clinical experiences as well as from case reports in the literature. The epidemiological study will determine the frequency of heterozygous mutations in the glucocerebrosidase gene and correlate to the clinical onset and development by measuring and documenting severity of symptoms (e.g. cognitive deficits, L-dopa responsiveness, depression) in clinically well-characterized Parkinson's patients.

DETAILED DESCRIPTION:
Parkinson's disease (also known as Parkinson's, Parkinson disease, or PD) is a degenerative disorder of the central nervous system that impairs motor skills, cognitive processes, and other functions. The most obvious symptoms are motor-related, including tremor, rigidity, slowness of movement, and postural instability. Among non-motor symptoms are autonomic dysfunction and sensory and sleep difficulties. Cognitive and neurobehavioral problems, including dementia, are common in the advanced stages of the disease. PD usually appears around the age of 60, although there are young-onset cases.

Gaucher's disease is a genetic disease in which a fatty substance (lipid) accumulates in cells and certain organs. Gaucher's disease is the most common of the lysosomal storage diseases. It is caused by a hereditary deficiency of the enzyme glucocerebrosidase (also known as acid β-glucosidase). The enzyme acts on a fatty substance glucocerebroside (also known as glucosylceramide). When the enzyme is defective, glucocerebroside accumulates, particularly in white blood cells (mononuclear leukocytes). Glucocerebroside can collect in the spleen, liver, kidneys, lungs, brain and bone marrow.

Symptoms of Parkinson's syndrome in classical type 1 Gaucher patients were first systematically described in 1996. In GD patients, a marked heterogeneity is detected in terms of disease-causing mutations. In 17 Gaucher patients with symptoms of Parkinson's disease, 12 different genotypes were sequenced and compared to other Parkinson's patients, a lower L-dopa responsiveness, a higher frequency of cortical dysfunction and a relatively early onset of the symptoms was described. Many of these Gaucher patients with clinical Parkinson's symptoms had a positive family history of Parkinson's disease among relatives with heterozygous mutations in the Gaucher gene that could be confirmed in systematic studies.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients at 18 years old
* Patients with confirmed diagnosis of Parkinson's disease
* Signed informed consent

Exclusion Criteria:

* Male or female patients being younger than 18 years old
* Patients without confirmed diagnosis of Parkinson's disease
* Missing signed informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adult patients with a confirmed diagnosis of Parkinson's disease
Sampling Method: Probability Sample
Enrollment: 1500 (Actual)
Dates: Start 2011-01 (Actual); Primary Completion 2016-06 (Actual); Study Completion 2017-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Arndt Rolfs, MD, Principal Investigator — University of Rostock, Albrecht-Kossel-Institute for Neuroregeneration
Locations (15):
- Germany (14):
  - Fachkrankenhaus für neurologische Akut- und Rehabilitationsmedizin, Bad Neustadt an der Saale
  - Universitätsklinikum Dresden Klinik für Neurologie, Dresden
  - University of Giessen, Department of Neurology, Giessen
  - Ernst-Moritz-Arndt-University of Greifswald, Department of Neurology, Greifswald
  - Universitätskrankenhaus Hamburg-Eppendorf, Department of Neurology, Hamburg
  - Medizinische Hochschule Hannover, Bewegungsstörungsambulanz, Hanover
  - Alexianer Krefeld GmbH, Krankenhaus Maria Hilf, Krefeld
  - Gertrudis-Kliniken im Parkinson-Zentrum, Leun
  - Neurologischische Arztpraxis, Rostock
  - Universitätsklinikum Rostock, Klinik für Neurologie, Rostock
  - Klinikverbund Südwest, Klinikum Sindelfingen-Böblingen, Sindelfingen
  - HANSE-Klinikum, Department of Neurology, Stralsund
  - University of Ulm, Department of Neurology, Ulm
  - Stiftung Deutsche Klinik für Diagnostik GmbH Fachbereich Neurologie, Wiesbaden
- Chulalongkorn University Hospital, Bangkok, Thailand

REFERENCES:
- [Background] Bras J, Singleton A, Cookson MR, Hardy J. Emerging pathways in genetic Parkinson's disease: Potential role of ceramide metabolism in Lewy body disease. FEBS J. 2008 Dec;275(23):5767-73. doi: 10.1111/j.1742-4658.2008.06709.x. PMID 19021754
- [Background] Clark LN, Ross BM, Wang Y, Mejia-Santana H, Harris J, Louis ED, Cote LJ, Andrews H, Fahn S, Waters C, Ford B, Frucht S, Ottman R, Marder K. Mutations in the glucocerebrosidase gene are associated with early-onset Parkinson disease. Neurology. 2007 Sep 18;69(12):1270-7. doi: 10.1212/01.wnl.0000276989.17578.02. PMID 17875915
- [Background] Gan-Or Z, Giladi N, Rozovski U, Shifrin C, Rosner S, Gurevich T, Bar-Shira A, Orr-Urtreger A. Genotype-phenotype correlations between GBA mutations and Parkinson disease risk and onset. Neurology. 2008 Jun 10;70(24):2277-83. doi: 10.1212/01.wnl.0000304039.11891.29. Epub 2008 Apr 23. PMID 18434642
- [Background] Goker-Alpan O, Schiffmann R, LaMarca ME, Nussbaum RL, McInerney-Leo A, Sidransky E. Parkinsonism among Gaucher disease carriers. J Med Genet. 2004 Dec;41(12):937-40. doi: 10.1136/jmg.2004.024455. PMID 15591280
- [Background] Kalinderi K, Bostantjopoulou S, Paisan-Ruiz C, Katsarou Z, Hardy J, Fidani L. Complete screening for glucocerebrosidase mutations in Parkinson disease patients from Greece. Neurosci Lett. 2009 Mar 13;452(2):87-9. doi: 10.1016/j.neulet.2009.01.029. Epub 2009 Jan 15. PMID 19383421
- [Background] Kitada T, Asakawa S, Hattori N, Matsumine H, Yamamura Y, Minoshima S, Yokochi M, Mizuno Y, Shimizu N. Mutations in the parkin gene cause autosomal recessive juvenile parkinsonism. Nature. 1998 Apr 9;392(6676):605-8. doi: 10.1038/33416. PMID 9560156
- [Background] Mitsui J, Mizuta I, Toyoda A, Ashida R, Takahashi Y, Goto J, Fukuda Y, Date H, Iwata A, Yamamoto M, Hattori N, Murata M, Toda T, Tsuji S. Mutations for Gaucher disease confer high susceptibility to Parkinson disease. Arch Neurol. 2009 May;66(5):571-6. doi: 10.1001/archneurol.2009.72. PMID 19433656
- [Background] Neudorfer O, Giladi N, Elstein D, Abrahamov A, Turezkite T, Aghai E, Reches A, Bembi B, Zimran A. Occurrence of Parkinson's syndrome in type I Gaucher disease. QJM. 1996 Sep;89(9):691-4. doi: 10.1093/qjmed/89.9.691. PMID 8917744
- [Background] Neumann J, Bras J, Deas E, O'Sullivan SS, Parkkinen L, Lachmann RH, Li A, Holton J, Guerreiro R, Paudel R, Segarane B, Singleton A, Lees A, Hardy J, Houlden H, Revesz T, Wood NW. Glucocerebrosidase mutations in clinical and pathologically proven Parkinson's disease. Brain. 2009 Jul;132(Pt 7):1783-94. doi: 10.1093/brain/awp044. Epub 2009 Mar 13. PMID 19286695
- [Background] Nichols WC, Pankratz N, Marek DK, Pauciulo MW, Elsaesser VE, Halter CA, Rudolph A, Wojcieszek J, Pfeiffer RF, Foroud T; Parkinson Study Group-PROGENI Investigators. Mutations in GBA are associated with familial Parkinson disease susceptibility and age at onset. Neurology. 2009 Jan 27;72(4):310-6. doi: 10.1212/01.wnl.0000327823.81237.d1. Epub 2008 Nov 5. PMID 18987351
- [Background] Sidransky E. Gaucher disease: complexity in a "simple" disorder. Mol Genet Metab. 2004 Sep-Oct;83(1-2):6-15. doi: 10.1016/j.ymgme.2004.08.015. PMID 15464415
- [Background] Sidransky E, Nalls MA, Aasly JO, Aharon-Peretz J, Annesi G, Barbosa ER, Bar-Shira A, Berg D, Bras J, Brice A, Chen CM, Clark LN, Condroyer C, De Marco EV, Durr A, Eblan MJ, Fahn S, Farrer MJ, Fung HC, Gan-Or Z, Gasser T, Gershoni-Baruch R, Giladi N, Griffith A, Gurevich T, Januario C, Kropp P, Lang AE, Lee-Chen GJ, Lesage S, Marder K, Mata IF, Mirelman A, Mitsui J, Mizuta I, Nicoletti G, Oliveira C, Ottman R, Orr-Urtreger A, Pereira LV, Quattrone A, Rogaeva E, Rolfs A, Rosenbaum H, Rozenberg R, Samii A, Samaddar T, Schulte C, Sharma M, Singleton A, Spitz M, Tan EK, Tayebi N, Toda T, Troiano AR, Tsuji S, Wittstock M, Wolfsberg TG, Wu YR, Zabetian CP, Zhao Y, Ziegler SG. Multicenter analysis of glucocerebrosidase mutations in Parkinson's disease. N Engl J Med. 2009 Oct 22;361(17):1651-61. doi: 10.1056/NEJMoa0901281. PMID 19846850
- [Background] Tayebi N, Walker J, Stubblefield B, Orvisky E, LaMarca ME, Wong K, Rosenbaum H, Schiffmann R, Bembi B, Sidransky E. Gaucher disease with parkinsonian manifestations: does glucocerebrosidase deficiency contribute to a vulnerability to parkinsonism? Mol Genet Metab. 2003 Jun;79(2):104-9. doi: 10.1016/s1096-7192(03)00071-4. PMID 12809640